CLINICAL TRIAL: NCT00305591
Title: Functional Magnetic Resonance Imaging and Spectroscopy of the Brain in Patients With Chronic Hepatic Encephalopathy
Brief Title: Brain Imaging in Patients With Chronic Liver Disease and Functional Impairment.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Royal College of Physicians (Other); Paddington Charitable Estates Educational Fund (Other); University of London (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 04/Q0406/161
Record Dates: First submitted 2006-03-21; First posted 2006-03-22 (Estimated); Last update posted 2015-05-29 (Estimated); Status verified 2008-01

CONDITIONS: Cirrhosis; Hepatic Encephalopathy
Keywords: magnetic resonance imaging; magnetic resonance spectroscopy; functional magnetic resonance imaging; cirrhosis; hepatic encephalopathy; l-ornithine l-aspartate
MeSH Terms: conditions — Fibrosis; Hepatic Encephalopathy | interventions — ornithylaspartate

INTERVENTIONS:
Drug: l-ornithine l-aspartate

SUMMARY:
Hepatic encephalopathy (HE) is a frequent complication of chronic liver disease (cirrhosis) and involves a wide spectrum of problems from mild impairment of reaction times in driving and operating machinery through to disturbances in mood, behaviour and conscious levels.

Magnetic resonance imaging (MRI) is a method of obtaining pictures of the inside of the body. Patients with liver disease have previously been studied with MRI which has highlighted changes in the brain. This research aims to highlight some of the differences in the way that the brain functions in patients with liver disease. Using our new, more powerful MRI scanner, with more sophisticated techniques we hope that the novel combination of MRI techniques can objectively detect the presence of , and monitor HE.

Study hypothesis: Hepatic encephalopathy (HE) is a reversible, metabolic disturbance of the brain, associated with low grade brain swelling and disturbances of the chemical balance within the brain, resulting in functional impairment, the presence of which MR imaging can detect with sufficient sensitivity to monitor the changes that may occur over time in response to treatment.

DETAILED DESCRIPTION:
Hepatic encephalopathy (HE) is a common neuropsychiatric abnormality, complicating the course of liver disease patients. In the UK, cirrhosis accounts for 4000 deaths per year, and 500,000 people are thought to be infected with chronic hepatitis C, of which up to 20% will develop cirrhosis over 20 years. The condition has been difficult to monitor objectively.

Despite the fact that the syndrome was probably first recognised two thousand years ago, the exact pathogenesis still remains unclear. It is thought to represent a reversible disturbance in brain chemistry and consequent brain swelling, in response to blood containing unfiltered gut-derived toxins entering the cerebral circulation. There is no recognised 'gold standard' test to diagnose and monitor this important, disabling condition. I have developed a novel combination of magnetic resonance imaging (MRI) sequences at 3 Tesla to study the effects of hepatic encephalopathy on the brain in patients with cirrhosis.

We propose to investigate alterations in brain size, function and chemistry before, and then at intervals after 4 weeks anti-encephalopathy treatment with L-ornithine L-aspartate. This will enable the assessment of both the baseline brain alterations of the cohort and the brain's response to therapy and correlation with their clinical response. As such this longitudinal study would allow us to define the sensitivity of the MR techniques.

Each of 50 patients will have blood tests, a 1 hour MRI brain scan and psychometric testing. The psychometric testing will be performed with both a computer-based battery and conventional paer-based tests. They will then be given L-ornithine L-aspartate (LOLA) to take orally for 4 weeks and have repeat blood tests, MRI and psychometric tests.

We will then determine if there is a correlation between the MR data and the results of the psychometric testing.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65
* Biopsy-proven cirrhosis
* Clinically stable
* Able to give informed consent
* Fluent English (required for psychometric testing)

Exclusion Criteria:

* Ferro-magnetic implants
* Claustrophobia
* Weight >120kg
* Significant renal impairment (Creatinine >150 micromol/L)
* Poorly controlled Diabetes (particularly type I with microvascular complications)
* Alcohol: if alcoholic liver disease is the aetiology of their liver disease they should be abstinent. Otherwise less than 20g per day.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2006-03; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
All enrolled patients will be given 4 weeks of treatment. Both MRI and functional changes will be observed.

CONTACTS AND LOCATIONS:
Overall Officials: Simon D Taylor-Robinson, MBBS, FRCP, Principal Investigator — Imperial College London & St Mary's Hospital
Locations (1):
- Imperial College London, Hammersmith, London, United Kingdom